CLINICAL TRIAL: NCT06306703
Title: Comparison of Teaching Methods of Pelvic Floor Muscle Contraction in Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duygu Sultan Oge (Other)
Responsible Party: Sponsor-Investigator, Duygu Sultan Oge, student, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PhD Thesis of Duygu Sultan Oge
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Pelvic Floor Muscle Weakness
Keywords: pelvic floor muscle contraction; pelvic floor assessment

STUDY DESIGN:
Intervention Model Description: prospective randomized
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: healthcare provider performing USG evaluation person doing statistical analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group1, verbal instruction (Experimental)
  Interventions: Other: group1, group2, group 3
- group 2, digital vaginal palpation (Experimental)
  Interventions: Other: group1, group2, group 3
- group 3, perineometer (Experimental)
  Interventions: Other: group1, group2, group 3

INTERVENTIONS:
Other: group1, group2, group 3 — to teaching with verbal instruction to teaching with digital vaginal palpation to teaching with perineometer

SUMMARY:
The aim of our study; To evaluate the effectiveness of different teaching methods on correct pelvic floor muscle contraction in women who have not received pelvic floor muscle training (PFMT) before. Women who come to the gynecology and obstetrics clinic for examination and volunteer for the study will be randomized with a computer-aided randomization program and divided into 3 groups. First of all, the pelvic floor muscles will be evaluated by ultrasonographic method and perineometer. The first group will be taught pelvic floor muscle contraction with verbal explanation, the second group will be taught with digital vaginal palpation, and the third group will be taught pelvic floor muscle contraction with the help of a perineometer. After the training, the same evaluations will be made again. The number of individuals to be included in the study will be determined by power analysis. As a result of this study, it will be decided which method can be used to teach pelvic floor muscle contraction to women accurately and effectively in clinics. The results of our study will guide clinicians in their preferences for using different teaching methods.

DETAILED DESCRIPTION:
The pelvic region, from inside to outside, consists of the endopelvic fascia that connects the pelvic organs to the side walls of the pelvis, the levator ani muscle (pubococcygeus, iliococcygeus and puborectalis), perineal membrane (urogenital diaphragm), external genital muscles (ischiocavernosus, bulbospongiosus and transversus perinei superficialis), external genital organs and It consists of skin. The perineal area is clinically the area between the vagina and the anus[1].

When the Levator Ani muscle was examined histochemically under an electron microscope, it was shown that it consisted of Type 1 (slow twitch-67%) and Type 2 (fast twitch-33%) striated muscle fibers. Type 1 fibers are resistant to fatigue and can produce contractions for long periods of time. Type 2 fibers have high contraction strength but have low resistance to fatigue. While Type 2 fibers cause sudden contraction in situations that increase intra-abdominal pressure, such as coughing, sneezing, heavy lifting, Type 1 fibers maintain the tone required for continence without fatigue for a long time [1, 2].

The pelvic floor has important functions in ensuring the continence mechanism, providing structural support to the pelvic openings such as the urethra, vagina and anus, supporting the pelvic organs, and performing vital activities such as sexual function and birth [3, 4].

Damage or weakening of the pelvic floor due to reasons such as pregnancy, birth, newborn weight, menopause, age, obesity, smoking, hysterectomy, constipation, systemic diseases, genetics, bad urination habits, constipation, heavy sports, or tension in the structures that form it. In this case, it may cause problems such as urinary incontinence, anorectal dysfunction, pelvic organ prolapse, pelvic pain or sexual dysfunction, and these pathologies are generally defined as pelvic floor dysfunction[4]. Although pelvic floor problems are not life-threatening, they affect people's psychological, social and physical well-being and negatively affect their quality of life by causing limitations in their work, family, social and sexual lives [5].

The pelvic floor can be evaluated by many different methods. The aim is to objectively evaluate the anatomy of the pelvic floor and pelvic organs and relate symptoms to anatomical findings. The methods used in the evaluation of the pelvic floor muscles are generally observation, palpation, electromyography (EMG), EMG with biofeedback, perineometer, pelvic floor dynamometer, ultrasonographic imaging (USG) and magnetic resonance imaging (MRI)[6]. Evaluations can be performed in the lithotomy position or standing.

There are two components to proper pelvic floor muscle contraction: compression of the pelvic openings and pulling inward in the cranial direction. Some explanations for why there is difficulty in voluntary pelvic floor muscle contraction: The fact that the pelvic floor muscles are in a place that cannot be seen in the pelvis, many people do not have knowledge about pelvic floor muscle contraction and are not aware of the automatic contractions of these muscles, from a neurophysiological point of view, voluntary contraction is difficult because the muscles are small, the pelvic and perineal areas are more prone to straining and defecation. and since they are related to excretion, the primary awareness is in this direction [7].

Some incorrect behaviors may occur while performing pelvic floor muscle contraction. These are reported as contraction of the abdominal muscles, hip adductor muscles or gluteal muscles instead of the pelvic floor muscles, holding the breath, excessive breathing and straining [7].

Studies in the literature report that more than 30% of women specifically have problems with pelvic floor muscle contraction [8]. There are studies reporting that approximately 25% of women perform the Valsalva maneuver instead when pelvic floor muscle contraction is requested [3]. In a study conducted in Austria, it was reported that during routine gynecological evaluation, 44.9% of women could not make correct pelvic floor muscle contraction and only 26.5% could perform muscle contraction without increasing intra-abdominal pressure [9]. There are studies reporting that when women contract their pelvic floor muscles, they also include other muscles in the contraction, and some of them strain their pelvic floor muscles rather than pulling them inwards [7]. In our study, investigators planned to evaluate the pelvic floor muscle contractions of women who had not received pelvic floor muscle training before and after different teaching methods and the compensations they used during this process.

Kegel reported that the majority of women did not have awareness of muscle function, so he performed the exercises with a perineometer, which makes muscle contraction visible with the help of an indicator. PTFE can be applied alone or using various devices such as biofeedback [8]. In our study, it was planned to teach one group only by verbal explanation, another group by digital vaginal palpation, and the third group by teaching pelvic floor muscle contraction with a perineometer.

In their study, Dietz et al. evaluated levator activity with transabdominal USG and aimed to teach patients levator muscle contraction directly on the screen by creating visual biofeedback with ultrasonography, with a maximum of 5 minutes of training. As a result, they emphasized that transabdominal USG provides good biofeedback to women who are not suitable for compensations and vaginal training. Thus, they advised women who came to the clinic for examination that pelvic floor muscle contraction could be taught in a very short time with USG [10]. In this study, based on this study, investigators will evaluate hiatal aperture and pelvic floor elevation with USG before and after different teaching methods.

Rodas et al. emphasize that pelvic floor muscle training should be specific to each patient and that the pelvic floor therapist should know which equipment or therapeutic aids are more effective to use for evaluation [2]. As a result of this study, investigators will discuss the advantages and disadvantages of pelvic floor muscle contraction teaching methods and provide clinicians with evidence-based information in this field.

In the literature, physiotherapy and rehabilitation approaches used to teach pelvic floor muscle contraction are verbal instructions, biofeedback, perineometer, vaginal cone, Foley catheter, tampon, three-dimensional real time ultrasound and virtual reality training. Verbal instructions used during training are necessary to elicit rapid and strong contraction of the pelvic floor muscles. One of the most frequently used verbal instructions in training is "Pinch and Pull" instruction. Another method for patients to understand correct pelvic floor muscle contraction is to use visual imagery techniques when describing the contraction. Visualizations such as closing the tap or door for squeezing, or the elevator going up for pulling in or holding can be used [7]. To describe correct muscle contraction, the movement can be likened to eating spaghetti, drinking water through a straw, the movement of a jellyfish, or the vacuum movement created in a vacuum cleaner. The investigator will use these metaphors in the training.

To the investigators knowledge, no study has been found in the literature comparing the techniques in which participants are taught pelvic floor muscle contraction with different methods before and after the training. The investigators think that will make new contributions to the literature in this field with their study.

ELIGIBILITY:
Inclusion Criteria:

* volunteering to participate in the study, getting a score of 25 or more from the "Mini mental Test", having pelvic floor muscle contraction ability, not having received pelvic floor muscle training before, vaginal examination and volunteering for education.

Exclusion Criteria:

* Pregnancy, presence of symptomatic pelvic organ prolapse over stage 2, cooperation problem, presence of urinary infection, epilepsy, and accompanying neurological disease.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 54 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
ASSESSMENT OF THE PELVIC FLOOR USING ULTRASONOGRAPHY (USG) | at the beginning 5 minutes, at the end 5 minutes
  During evaluation with 2D USG, hiatal aperture measurements will be made at rest and at maximum voluntary contraction. Measurements will be repeated before and after individuals receive training, and any numerical changes that may occur will be recorded[11,12].
Pelvic Floor Muscle Strength and Endurance: | 5 minutes
  Pelvic floor muscle strength and endurance will be evaluated with a non-invasive vaginal perineometer with digital vaginal palpation
pelvic floor power, minimum and maximum muscle contraction values | 5 minutes
  Pelvic floor power will be evaluated with intravajinal biofeedback electromyograhy(EMG)

SECONDARY OUTCOMES:
DETAILED STORIES OF THE PATIENTS | 5 minutes
  The physical characteristics of the patients such as age (years), height, weight, BMI, demographic data such as educational status, employment status, and marital status will be recorded. The detailed history will include a CV inquiring about chronic diseases and surgeries, a family history inquiring about diseases in first-degree relatives, and a gynecological history inquiring about previous gynecological diseases and surgeries, if any. The patients' obstetric history, which questions gravida (number of pregnancies), parity (number of births), abortus (number of miscarriages), number of dilations and curettages, type of birth, birth weight and interventions used at birth, will also be recorded. In addition; Menstrual status (regular menstruation, irregular menopause, spontaneous menopause, surgical menopause) will be questioned.
Pelvic Floor Health Knowledge Test: | 5 minutes
  This test, developed and validated by Al-Deges et al., consists of 29 questions. The 'test yes-no-don't know?' which contains questions about pelvic floor health. It is answered with options. This test will be applied to women before they receive pelvic floor training. In this way, the knowledge level of the women included in the study about the pelvic floor will be evaluated[13].
Global Pelvic Floor Disorder Questionnaire(GPFDQ) | 5 minutes
  GPFDQ, which is used in the evaluation and determination of the severity of stress urinary incontinence, frequent urination, sudden urination, urge incontinence, urination difficulty, pelvic organ prolapse, obstructive defecation, anal incontinence and dyspareunia symptoms, which are frequently encountered in pelvic floor dysfunctions, has been adapted to Turkish, its validity and It is a reliable survey. In our study, we will use this survey to eliminate women's discomfort regarding these problems [14].
Visual Analog Scale (VAS) assessment for pelvic pain | 1 minute
  VAS scores will be recorded to question the pelvic pain of the women included in the study. In the 10-centimeter long VAS, 0 indicates no pain, while 10 indicates the most severe pain. Individuals are asked to mark the part on the scale that expresses their pain [15].
Determining the severity of incontinence | 1 minute
  The International Incontinence Severity Index is used to reveal the severity, frequency and type of urinary incontinence and to show how much urinary incontinence affects the person's quality of life[16].
Sensory Evaluation | 1 minute
  Sensory test will be performed as a result of sharp-blunt, hot-cold tests applied to the sensory area innervated by the sacral 2-4 segmental nerves, in order to determine whether the patient has any sensory loss in these dermatomes [17].
Pelvic Floor Reflex Evaluation: | 1 minute
  As part of the neurological examination, evaluation of the pudendal nerve and Sacral 2-4 sacral reflexes should be performed. In evaluating the bulbocavernous reflex, a cotton swab will be passed over the labia minora to check whether both labia contract equally. Secondly, in the anal reflex, the contraction caused by rubbing the cotton swab against the perianal skin will be evaluated[18].
Evaluation of Mistakes Made During Pelvic Floor Muscle Contraction | 5 minutes
  Contraction of abdominal muscles instead of pelvic floor muscles: While the evaluations are being made, biofeedback EMG (NeuroTrac® Myo Plus Pro) superficial electrodes will be placed at the spina iliaca anterior superiors level for possible contraction in the abdominal muscles and the muscle activation response will be recorded in mV..
  Contraction of adductor muscles instead of pelvic floor muscles, Contraction of the gluteal muscles instead of the pelvic floor muscles, Excessive breathing, Holding the breath and pushing(7).
Pelvic organ prolapse evaluation | 1 minute
  to classified pelvic organ prolapse

CONTACTS AND LOCATIONS:
Overall Officials: Türkan Akbayrak, Prof, Study Director — Hacettepe Universty

IPD SHARING:
Plan to Share IPD: No